CLINICAL TRIAL: NCT06215131
Title: Feasibility of Immersive Virtual Reality Dietician Program in Patients With Metabolic-dysfunction Associated Steatotic Liver Disease
Brief Title: Feasibility of Immersive Virtual Reality Dietician Program in Metabolic-dysfunction Associated Steatotic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Justin Tondt, Assistant Professor of Family and Community Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00024998
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Fatty Liver, Nonalcoholic; Weight Loss; Virtual Reality; Implementation Science
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person dietary weight loss counseling (Active Comparator): The counseling content will be 30 minutes of RDN delivered educational session on energy density and portion sizes then the second 30 minutes being the RDN answering participant questions and providing feedback.
  Interventions: Behavioral: In-person dietary weight loss counseling
- Virtual reality dietary weight loss counseling (Experimental): The counseling content will be 30 minutes of virtual reality delivered educational session on energy density and portion sizes with an RDN remotely monitoring then the second 30 minutes being the RDN answering participant questions and providing feedback through synchronous audio/video.
  Interventions: Behavioral: Virtual reality dietary weight loss counseling

INTERVENTIONS:
Behavioral: In-person dietary weight loss counseling — The counseling content will be 30 minutes of RDN delivered educational session on energy density and portion sizes then the second 30 minutes being the RDN answering participant questions and providing feedback.
  Arms: In-person dietary weight loss counseling
Behavioral: Virtual reality dietary weight loss counseling — The counseling content will be 30 minutes of virtual reality delivered educational session on energy density and portion sizes with an RDN remotely monitoring then the second 30 minutes being the RDN answering participant questions and providing feedback through synchronous audio/video.
  Arms: Virtual reality dietary weight loss counseling

SUMMARY:
Metabolic-dysfunction associated steatotic liver disease, often referred to as "fatty liver disease", is a leading cause of liver failure. Dietary weight loss is a cornerstone of treating fatty liver disease, but access to traditional in-person nutritional education is often limited by cost, availability, and transportation. Immersive virtual reality (iVR) has the potential to not only overcome these barriers, but also provide an interactive learning experience, such as measuring and preparing foods. Therefore, the investigators have created and validated an iVR dietician program known as the Immersive Virtual Alimentation and Nutrition (IVAN) using evidence-informed practices from the Academy of Nutrition and Dietetics.

The goal of this project is to translate the IVAN program from human and patient research to practice and community research. The investigators plan to accomplish this by performing a randomized clinical trial evaluating the effect of the IVAN program in combination with synchronous audio/video dietary counseling on self-reported dietary intake and weight compared to in-person counseling. Concurrently, the investigators will provide a survey assessing implementation outcomes to both groups as well as the dietician at each study visit, and crossover the intervention at study completion so all participants assess the IVAN program. Additionally, the investigators will have clinic health care providers experience the IVAN program and assess implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >18 years
* MASLD identified on imaging
* Possession of a smartphone

Exclusion Criteria:

* Inability to provide informed consent
* Institutionalized/prisoner
* Pregnant
* Other causes of hepatic steatosis or chronic liver disease
* Severe medical/psychiatric comorbidities at the study PI's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Kg
Change in percent body weight | 12 weeks
  Percent change

SECONDARY OUTCOMES:
Change in energy intake | 12 weeks
  Calories via ASA24
Change in hepatic steatosis | 12 weeks
  Liver fat measured via Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Justin Tondt, MD, Principal Investigator — Penn State
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No